CLINICAL TRIAL: NCT04947332
Title: Effectiveness of Auto-inoculation of a Wart in Multiple Viral Warts, in Tertiary Care Hospital : A Single Arm Study
Brief Title: Auto-inoculation of a Wart in Multiple Viral Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pak Emirates Military Hospital (Other)
Responsible Party: Principal Investigator, Muhammad Waseem Shahid, Resident Dermatology, Pak Emirates Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A/28/EC/230/2021
Record Dates: First submitted 2021-06-19; First posted 2021-07-01 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Viral Wart; Delayed Hypersensitivity
Keywords: Autoinoculation; Viral Warts; Hypersensitivity; Immunology
MeSH Terms: conditions — Warts; Hypersensitivity, Delayed; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: A single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auto-inoculation recipients (Other): Auto-inoculation of wart to be performed
  Interventions: Procedure: Auto-inoculation

INTERVENTIONS:
Procedure: Auto-inoculation — A wart will be excised from the body, minced and will be inoculated in a subcutaneous pocket on forearm.

SUMMARY:
This study is being conducted to see effectiveness of auto-inoculation of a wart in multiple viral warts. Patients with recurrent, multiple warts of all types, are being recruited for the study. A wart is excised, minced and then inoculated in a subcutaneous pocket made on the volar aspect of forearm. Patients are to be reviewed after every 4 weeks to note any reduction in number warts.

DETAILED DESCRIPTION:
A single arm, Phase 1, Clinical Study

ELIGIBILITY:
Inclusion Criteria:

* Individuals having 5 or warts
* Individuals having any types of warts

Exclusion Criteria:

* Individuals using any other treatment for warts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
Complete Clearance of Warts | 12 weeks
  All the warts on any part of the body are cleared
Incomlete Clearance of Warts | 12 weeks
  No or size of warts are reduced
Non Responders | 12 weeks
  If no change or increased no of warts

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Iftikhar, MBBS, FCPS, Study Director — Head of Department
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No